CLINICAL TRIAL: NCT01130220
Title: Informed Brain Cancer Patients
Brief Title: Study of the Health Information Needs of Brain Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 708-2009
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Focus Groups

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Brain Tumor Patient: A one-time focus group will be held in a quiet room for approximately 30-60 minutes until a "saturation" of themes has been identified.
  Interventions: Other: Focus Group
- Health Care Provider: A one-time focus group will be held in a quiet room for approximately 30-60 minutes until a "saturation" of themes has been identified.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — A single focus group will be held until a "saturation" of themes has been identified.

SUMMARY:
The purpose of this research is to explore the factors involved in brain cancer health care literacy needs.

DETAILED DESCRIPTION:
A mere subset of the reasons behind unmet health care literacy needs include the health care systems' increasing complexity, increased time constraints, profound treatment decision making requirements, decreased financial resources, fracturing social networks and diversifying educational and cultural needs.

This project will use focus groups to explore the factors involved in brain cancer health care literacy from the perspectives of patients and those involved in their care. Hypothesis generated from this project will be directly applied toward future projects. The overarching goals are improved access and adequacy of health care literacy information through the eventual development of validated, useful, reliable health care literacy information tools for brain cancer patients and those involved in their care.

ELIGIBILITY:
Inclusion Criteria:

BRAIN TUMOR PATIENTS:

* 18 to 89 years of age
* Have or have had any type of brain tumor
* Ability to communicate in English
* Willingness to participate in a 30-60 minute focus group

HEALTH CARE PROVIDERS:

* 18 to 89 years of age
* Be a health care provider who cares for any type of brain tumor
* Ability to communicate in English
* Willingness to participate in a 30-60 minute focus group

Exclusion Criteria:

* None

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited during routine interactions with the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Explore the factors involved in health care literacy from the perspective of brain cancer patients. | 1 Year
  An investigator experienced in semi-structured focus group research will faclitate focus group sessions by using a generalized list of topics and open-ended discussion questions.

SECONDARY OUTCOMES:
Explore the factors involved in health care literacy from the perspective of health care providers. | 1 Year
  An investigator experienced in semi-structured focus group research will faclitate focus group sessions by using a generalized list of topics and open-ended discussion questions.

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Dunbar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States